CLINICAL TRIAL: NCT04201392
Title: Prevalence and Characteristics of Sleep Disturbances Among Psychiatric Inpatients
Brief Title: Sleep in Psychiatric Inpatients
Acronym: SPIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01297
Record Dates: First submitted 2019-10-03; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Sleep Disturbance; Sleep Disorder; Insomnia; Hypersomnia; Psychiatric Disorder
Keywords: Psychiatric inpatient care
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Decades of research have shown that sleep disturbances are common among patients with a wide range of psychiatric disorders. Such reported sleep disturbances include disrupted sleep efficiency and continuity, sleep quality complaints, insomnia, and nightmares. While traditional models suggest that certain sleep alterations are specific for certain mental disorders, newer models assume a transdiagnostic or dimensional view of sleep disturbances in mental disorders. Findings of a recent meta-analysis support the transdiagnostic or dimensional association between sleep disorders and psychiatric conditions. Additionally, the period just prior to sleep has recently received increased clinical and research interest, with studies investigating cognitive activity and rumination prior to sleep. However, only few studies compare sleep in different psychiatric diagnoses and the characteristics of sleep in different mental disorders are still not understood well enough for concrete implications for clinical practice. This is especially true for the population of psychiatric inpatients. In this study, the outcome measures and study variables will be measured with standardised and validated questionnaires, structured clinical interview, and a commercially available Fitbit Charge 2 tracker. Participants will be recruited from the inpatient units of the Psychiatric University Hospital Zurich (PUK). Screening will be conducted by the applicant and master's students enrolled in the project, using electronic patient files at the hospital. The patients will be invited to the study by their treating physician or psychologist. Assessments will consist of one interview and filling out of questionnaires (with a 30- to 45-minute duration respectively). A sub-sample will wear fill out a sleep diary for seven consecutive nights as well as wear a Fitbit Charge 2 tracker, which they will return a week later. Each patient will receive participant reimbursement of 30 Swiss francs (CHF) for their participation in the study.

DETAILED DESCRIPTION:
Sleep disturbances are common among psychiatric patients. In fact, most psychiatric disorders are afflicted with sleep disturbances. Mechanistical underpinnings and associations between sleep disturbances and psychiatric conditions have been an active field of research. Individuals with alcohol or substance abuse reported disrupted sleep efficiency and continuity, as well as rates of insomnia as high as 72%. In schizophrenia, insomnia and other sleep-related abnormalities are also common, with prevalence rates of 30% to 80%. Moreover, individuals with mood disorders describe a range of difficulties with sleep continuity and quality. Another study in depressed individuals reported rates as high as 90% of reported sleep quality complaints. Similarly, anxiety disorders are highly associated with sleep disorders. The fact that sleep disturbance is a diagnostic symptom for disorders such as generalized anxiety disorder and post-traumatic stress disorder (PTSD) underpins the relationship between anxiety and sleep. In PTSD for example, difficulty initiating and maintaining sleep and nightmares affect approximately 70% of individuals afflicted with this disorder. Reexperiencing in the form of distressing dreams and intrusive trauma memories prior to initiating sleep are commonly reported in this group. Taken together, these reports show that sleep problems are common in psychiatric patients. Some theoretical models suggest that certain sleep alterations are specific for certain mental disorders. Newer models, however, suggest a transdiagnostic or dimensional understanding of sleep in mental disorders, assuming sleep as an underlying dimension of mental disorders, with the same sleep alterations occurring in different mental disorders. Few studies comprise large enough numbers to compare different psychiatric diagnoses, however, and thus, few data exist on the specificity of various sleep abnormalities. In a notable exception, a meta-analysis investigated sleep disturbances across psychiatric disorders, reviewing studies using polysomnographic measurements. The authors found that no single sleep variable appeared to have absolute specificity for any particular psychiatric disorder and that patterns of sleep disturbances associated with categories of psychiatric disorders were observed. Additionally, the subtypes of diagnosis groups often differed in their profiles of sleep alterations. Thus, these results support the transdiagnostic view of sleep disturbances in mental disorders. In the light of these findings, however, it is interesting that the period just prior to sleep onset has recently received increased research and clinical interest. Pre-sleep cognitive activity of individuals suffering from insomnia has been shown to be more focused on worries, problems and noises in the environment and less focused on nothing in particular, compared to good sleepers. There is also evidence that rumination prior to sleep is associated with sleep disturbance (increased sleep onset latency, reduced sleep quality, reduced sleep efficiency, and increased wakefulness after sleep onset). Identification of potential disorder-specific as well as transdiagnostic pre-sleep processes would be helpful for diagnosing and treating patients. This is particularly important considering the heavy personal burden associated with psychiatric disorders and sleep disturbances. Most of the studies investigating sleep disturbances in psychiatric disorders have been conducted in psychiatric outpatients. Psychiatric inpatients and the even more severely afflicted patients who often suffer from comorbid diagnoses and possible additional social problems, have so far been mostly excluded. There are a few studies, which investigated sleep problems in psychiatric inpatients and/or patients with severe mental illness. Furthermore, although the period just prior to sleep onset has recently received increased research and clinical interest, a systematic investigation of individuals with diagnosed psychiatric disorders in terms of this specific sleep characteristic is lacking so far. The present study therefore aims to help fill this gap and study sleep problems, including pre-sleep processing in psychiatric inpatients. Additionally, studies investigating sleep disturbances using samples of patients with different psychiatric disorders are lacking. Thus, in order to understand the differences in sleep disturbances between different psychiatric diagnoses or symptom clusters, different studies have to be compared. Since these studies often differ in the samples and methods used, conclusions drawn from these comparisons are limited. For this reason, studies using samples of psychiatric patients with a wide range of psychiatric disorders are warranted.

For this study, participants will be recruited from the inpatient units of the Psychiatric University Hospital Zurich (PUK). Consultant psychiatrists and psychologists, as well as nursing personnel in the inpatient units of the PUK will support recruitment and one or two master students will help organise the study. All patients eligible for the study will be recruited consecutively. The applicant and master's students enrolled in the project will screen newly admitted psychiatric inpatients for inclusion and exclusion criteria in the electronic patient files. The information needed for the screening is part of standard assessments at the hospital. The treating psychologists or physicians will then be contacted directly by the applicant or master's students. The treating psychologists and physicians will invite the patients who meet the inclusion and exclusion criteria to the study. Prior to the first session, the applicant or master's students will use the patient's electronic file to document medical information, such as medical history, current primary diagnosis, and current medication. The first session, which will be led by the applicant or master's students, will consist of informed consent, a clinical interview, and a first set of self-report questionnaires, which will assess primary psychiatric diagnoses, measure demographic and personal information, sleep disorders, sleep characteristics, several psychological variables (such as emotional regulation, rumination, and mindfulness) and current symptom severity of the primary diagnosis. A sub-sample of patients will receive a sleep diary and a Fitbit Charge 2 tracker as well as information regarding its application. They will wear the Fitbit tracker on the wrist of their non-dominant hand at all times for a week (except during showers and / or charging). A week later, the questionnaires and/or diary and Fitbit tracker will be collected. Additionally, patients will be asked if they have any questions or whether they ran into any problems. After data collection is completed, each patient will receive participant reimbursement of 30 Swiss francs (CHF) for their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients from PUK inpatient units between 18 and 65 years of age
* ICD-10 diagnosis of affective disorders (F32, F33, F34.1), substance use disorders (F10.2, F12.2, F14.2), anxiety disorders (F40.0, F40.1, F40.2, F41.0, F41.1), and schizophrenia (F20.0)
* Currently receiving inpatient care at the Psychiatric University Hospital Zurich
* Fluent in German and able to understand the instructions

Exclusion Criteria:

* Currently receiving outpatient or day clinic programs at the Psychiatric University Hospital Zurich
* ICD-10 diagnosis other than F32, F33, F34.1, F10.2, F12.2, F14.2, F40.0, F40.1, F40.2, F41.0, F41.1, and F20.0
* Patients who are too severely ill to fill in questionnaires
* Patients with a one on one or 15- / 30-minute visual control by the nursing personnel because of risk of suicidal tendencies or the risk of harming others
* Head injury
* Neurological disease
* Shift work
* Trouble speaking and / or understanding German language

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For this study, participants will be recruited from the inpatient units at the Psychiatric University Hospital Zurich (PUK). It is aimed to recruit patients from each of the following diagnostic groups: Affective disorders, substance use disorders, anxiety disorders, and schizophrenia. These groups have been chosen, because they are the biggest patient groups in the hospital. Within the groups, the most common diagnoses among inpatients at the PUK will be investigated (F32, F33, F34.1, F10.2, F12.2, F14.2, F40.0, F40.1, F40.2, F41.0, F41.1, and F20.0). A sub-sample from the same sample will be recruited for Fitbit tracker measurements. Participation in the research will be fully independent of their treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep disorders | 7 days
  The Sleep Disorders Symptom Checklist and the sleep module of the Diagnostische Interview bei psychischen Störungen will measure current sleep disorders as listed in the DSM-IV-TR and DSM-V (sleep apnea, insomnia, narcolepsy, restless legs/PLMD, circadian rhythm sleep disorder, sleepwalking, nightmares, factors influencing sleep, and the impact of sleep complaints on daily functioning).
Characteristics of sleep disturbances: Subjective total sleep time | 7 days
  The Pittsburg Sleep Quality Index and the sleep module of the Diagnostische Interview bei psychischen Störungen will measure current subjective total sleep time.
Characteristics of sleep disturbances: Objective total sleep time | 7 days
  The Fitbit Charge 2 will measure daily objective total sleep time.
Characteristics of sleep disturbances: Subjective sleep onset latency | 7 days
  The Pittsburg Sleep Quality Index and the sleep module of the Diagnostische Interview bei psychischen Störungen will measure current subjective sleep onset latency.
Characteristics of sleep disturbances: Objective sleep onset latency | 7 days
  The Fitbit Charge 2 will measure daily objective sleep onset latency.
Characteristics of sleep disturbances: Subjective wake after sleep onset | 7 days
  The Pittsburg Sleep Quality Index and the sleep module of the Diagnostische Interview bei psychischen Störungen will measure current minutes awake after sleep onset.
Characteristics of sleep disturbances: Objective wake after sleep onset | 7 days
  The Fitbit Charge 2 will measure daily minutes awake after sleep onset.
Characteristics of sleep disturbances: Daily subjective total sleep time | 7 days
  A sleep diary will measure daily subjective total sleep time.
Characteristics of sleep disturbances: Daily subjective sleep onset latency | 7 days
  A sleep diary will measure daily subjective sleep onset latency.
Characteristics of sleep disturbances: Daily subjective wake after sleep onset | 7 days
  A sleep diary will measure minutes awake after sleep onset for each night.
Characteristics of sleep disturbances: Subjective sleep quality | 7 days
  The Pittsburg Sleep Quality Index will measure current sleep quality. Higher Pittsburgh Sleep Quality Index scores indicate lower sleep quality (minimum value: 0, maximum value: 21).
Characteristics of sleep disturbances: Daytime sleepiness | 7 days
  Daytime sleepiness will be measured specifically by the Epworth Sleepiness Scale (minimum value: 0, maximum value: 24).
Characteristics of sleep disturbances: Subjective sleep efficiency | 7 days
  The Pittsburg Sleep Quality Index will measure current subjective sleep efficiency.
Characteristics of sleep disturbances: Chronotype | 7 days
  The Munich Chronotype Questionnaire will measure chronotype based on the midpoint of a person's sleep.
Characteristics of sleep disturbances: Dream experiences and believes | 7 days
  The Mannheim Dream Questionnaire will measure dream experiences and believes.
Characteristics of sleep disturbances: Nightmare frequency | 7 days
  The Mannheim Dream Questionnaire will measure current nightmare frequency.
Characteristics of sleep disturbances: Nightmare distress | 7 days
  The Mannheim Dream Questionnaire will measure nightmare distress.
Characteristics of sleep disturbances: Daily nightmare frequency | 7 days
  A sleep diary will measure daily prospective nightmare frequency.
Characteristics of sleep disturbances: Daily nightmare distress | 7 days
  A sleep diary will measure daily prospective nightmare distress.
Characteristics of sleep disturbances: Heart rate during sleep | 7 days
  A Fitbit device will measure average heart rate (bpm) during sleep.
Processes of psychopathology other than sleep: Trait mindfulness | 7 days
  The Mindful Attention Awareness Scale will measure current trait mindfulness. Higher Mindful Attention Awareness Scale scores indicate higher trait mindfulness (minimum value: 15, maximum value: 90).
Processes of psychopathology other than sleep: State mindfulness | 7 days
  A sleep diary will measure daily state mindfulness.
Processes of psychopathology other than sleep: Trait rumination | 7 days
  The Response Styles Questionnaire will measure trait rumination. Higher Response Styles Questionnaire scores indicate higher trait rumination, divided into a brooding and a reflection score (minimum brooding and reflection values: 5, maximum brooding and reflection values: 20).
Processes of psychopathology other than sleep: State rumination | 7 days
  A sleep diary will measure daily state rumination.
Processes of psychopathology other than sleep: Emotional regulation | 7 days
  The Emotion Regulation Questionnaire will measure emotional regulation divided into two emotion regulation processes: Reappraisal and suppression. Higher values indicate higher tendencies for reappraisal (minimum value: 6, maximum value: 42) or suppression (minimum value: 4, maximum value: 28).

SECONDARY OUTCOMES:
Psychiatric diagnosis | 1 day
  The Mini International Neuropsychiatric Interview is a diagnostic interview, which will measure, which psychiatric diagnosis / diagnoses are met according to the International Classification of Diseases (ICD-10) and the Diagnostic and Statistical Manual of Mental Disorders (DSM 4).
Current severity of depressive symptoms | 7 days
  The Beck Depression Inventory will measure current severity of depressive symptoms (minimum value: 0, maximum value: 63). Higher scores indicate a higher severity.
Current severity of anxiety symptoms | 7 days
  The Beck Anxiety Inventory will measure current severity of anxiety symptoms (minimum value: 0, maximum value: 63). Higher scores indicate a higher severity.
Current severity of alcohol use | 7 days
  The Alcohol Use Disorders Identification Test will measure current severity of alcohol use (minimum value: 0, maximum value: 40). Higher scores indicate a higher severity.
Current severity of drug use | 7 days
  The Drug Use Disorders Identification Test will measure current severity of drug use (minimum value: 0, maximum value: 44). Higher scores indicate a higher severity.
Current severity of PTSD symptoms | 7 days
  The PTSD Checklist for DSM-5 will measure current severity of PTSD symptoms (minimum value: 0, maximum value: 80). Higher scores indicate a higher severity.
Current severity of psychotic symptoms | 7 days
  The Community Assessment of Psychic Experiences will measure current severity of psychotic symptoms (frequency and distress score with minimum value: 0, maximum value: 126). Higher scores indicate a higher severity.
Current severity of schizophrenia symptoms | 7 days
  The Positive and Negative Syndrom Scale will measure current severity of schizophrenia symptoms (minimum value: 30, maximum value: 210). Higher scores indicate a higher severity.

OTHER OUTCOMES:
Demographic and personal information | 7 days
  A questionnaire will measure demographic and medical background information, such as sex, age, nationality, marital status, residence permit status, children, life situation, highest education, current or last work situation, current social situation, socioeconomic status.
Current medication | 7 days
  As a potential confounder, a medication protocol will measure current medication, especially medication, which has been reported to have an effect on sleep, will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rumble ME, White KH, Benca RM. Sleep Disturbances in Mood Disorders. Psychiatr Clin North Am. 2015 Dec;38(4):743-59. doi: 10.1016/j.psc.2015.07.006. PMID 26600106
- [Background] Ford DE, Kamerow DB. Epidemiologic study of sleep disturbances and psychiatric disorders. An opportunity for prevention? JAMA. 1989 Sep 15;262(11):1479-84. doi: 10.1001/jama.262.11.1479. PMID 2769898
- [Background] Benca RM, Obermeyer WH, Thisted RA, Gillin JC. Sleep and psychiatric disorders. A meta-analysis. Arch Gen Psychiatry. 1992 Aug;49(8):651-68; discussion 669-70. doi: 10.1001/archpsyc.1992.01820080059010. PMID 1386215
- [Background] Krystal AD, Thakur M, Roth T. Sleep disturbance in psychiatric disorders: effects on function and quality of life in mood disorders, alcoholism, and schizophrenia. Ann Clin Psychiatry. 2008 Jan-Mar;20(1):39-46. doi: 10.1080/10401230701844661. PMID 18297585
- [Background] Baglioni C, Nanovska S, Regen W, Spiegelhalder K, Feige B, Nissen C, Reynolds CF, Riemann D. Sleep and mental disorders: A meta-analysis of polysomnographic research. Psychol Bull. 2016 Sep;142(9):969-990. doi: 10.1037/bul0000053. Epub 2016 Jul 14. PMID 27416139
- [Background] Harvey AG. Pre-sleep cognitive activity: a comparison of sleep-onset insomniacs and good sleepers. Br J Clin Psychol. 2000 Sep;39(3):275-86. doi: 10.1348/014466500163284. PMID 11033749
- [Background] Thomsen, D. K., Mehlsen, M. Y., Christensen, S., & Zachariae, R. (2003). Rumination: Relationship with negative mood and sleep quality, Personality and Individual Differences, 34(7), 1293-1301. doi: 10.1016/S0191-8869(02)00120-4
- [Background] Takano K, Iijima Y, Tanno Y. Repetitive thought and self-reported sleep disturbance. Behav Ther. 2012 Dec;43(4):779-89. doi: 10.1016/j.beth.2012.04.002. Epub 2012 Apr 19. PMID 23046780
- [Background] Carney CE, Edinger JD, Meyer B, Lindman L, Istre T. Symptom-focused rumination and sleep disturbance. Behav Sleep Med. 2006;4(4):228-41. doi: 10.1207/s15402010bsm0404_3. PMID 17083303
- [Background] Carney CE, Harris AL, Moss TG, Edinger JD. Distinguishing rumination from worry in clinical insomnia. Behav Res Ther. 2010 Jun;48(6):540-6. doi: 10.1016/j.brat.2010.03.004. Epub 2010 Mar 11. PMID 20362977
- [Background] Roehrs, T., & Roth, T. (2012). Sleep and sleep disorders. In J. C. Verster, K. Brady, M. Galanter, & P. Conrod (Eds.), Drug abuse and addiction in medical illness: Causes, consequences and treatment (S. 375-384). New York: Springer Science + Business Media.
- [Background] Kamath J, Virdi S, Winokur A. Sleep Disturbances in Schizophrenia. Psychiatr Clin North Am. 2015 Dec;38(4):777-92. doi: 10.1016/j.psc.2015.07.007. Epub 2015 Aug 22. PMID 26600108
- [Background] Tsuno N, Besset A, Ritchie K. Sleep and depression. J Clin Psychiatry. 2005 Oct;66(10):1254-69. doi: 10.4088/jcp.v66n1008. PMID 16259539
- [Background] Staner L. Sleep and anxiety disorders. Dialogues Clin Neurosci. 2003 Sep;5(3):249-58. doi: 10.31887/DCNS.2003.5.3/lstaner. PMID 22033804
- [Background] Ohayon MM, Shapiro CM. Sleep disturbances and psychiatric disorders associated with posttraumatic stress disorder in the general population. Compr Psychiatry. 2000 Nov-Dec;41(6):469-78. doi: 10.1053/comp.2000.16568. PMID 11086154
- [Background] Nappi CM, Drummond SP, Hall JM. Treating nightmares and insomnia in posttraumatic stress disorder: a review of current evidence. Neuropharmacology. 2012 Feb;62(2):576-85. doi: 10.1016/j.neuropharm.2011.02.029. Epub 2011 Mar 17. PMID 21396945
- [Background] Babson K, Feldner M, Badour C, Trainor C, Blumenthal H, Sachs-Ericsson N, Schmidt N. Posttraumatic stress and sleep: differential relations across types of symptoms and sleep problems. J Anxiety Disord. 2011 Jun;25(5):706-13. doi: 10.1016/j.janxdis.2011.03.007. Epub 2011 Mar 17. PMID 21482065
- [Background] Harvey AG, Jones C, Schmidt DA. Sleep and posttraumatic stress disorder: a review. Clin Psychol Rev. 2003 May;23(3):377-407. doi: 10.1016/s0272-7358(03)00032-1. PMID 12729678
- [Background] Mume, C. O. (2009). Nightmare in schizophrenic and depressed patients, European Journal of Psychiatry, 23(3), 177-183.
- [Background] Kaufmann CN, Spira AP, Rae DS, West JC, Mojtabai R. Sleep problems, psychiatric hospitalization, and emergency department use among psychiatric patients with Medicaid. Psychiatr Serv. 2011 Sep;62(9):1101-5. doi: 10.1176/appi.ps.62.9.1101. PMID 21885593